CLINICAL TRIAL: NCT02328690
Title: Binaural Beat Technology: A Complementary Path to Post Deployment Wellness (The Sound Mind Warrior Study)
Brief Title: The Sound Mind Warrior Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fort Belvoir Community Hospital (U.S. Federal Agency)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); TriService Nursing Research Program (Other)
Responsible Party: Principal Investigator, LTC MeLisa Gantt, (former) Chief, Research Program, Fort Belvoir Community Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 361395
Record Dates: First submitted 2014-12-18; First posted 2014-12-31 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Anxiety; Stress
Keywords: binaural beat technology; sound technology; cardiovascular stress response; military; music; anxiety; stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music with BBT (Experimental): Music embedded with special tones.
  Interventions: Other: Binaural Beat Technology
- Music without BBT (Placebo Comparator): Music not embedded with special tones.
  Interventions: Other: Binaural Beat Technology

INTERVENTIONS:
Other: Binaural Beat Technology — A phenomenon when two nearly similar frequencies (between 30-1000 hertz [Hz]) are presented to each ear and the brain detects the difference between the two sounds. These two sounds are processed in the superior olivary nucleus of each hemisphere of the brain. This integration of brain hemispheres produces a frequency that in turn affects the reticular activating system which alters the electrical potentials of the thalamus and cerebral cortex changing brainwave frequency.
  Other Names: Hemi-Sync

SUMMARY:
The purpose of this prospective, double-blind, repeated measures study is to assess the efficacy of Binaural Beat Technology (BBT) on anxiety and anxiety related cardiovascular measures as well as to assess the feasibility of implementing a BBT intervention in a military population during the high risk post-deployment window.

DETAILED DESCRIPTION:
The purpose of this prospective, double-blind, repeated measures study is to assess the efficacy of Binaural Beat Technology (BBT- a sound technology that uses special tones [embedded in music] through stereo headphones to affect your brainwaves in order to put you in a more relaxed state) on anxiety and anxiety related cardiovascular measures as well as to assess the feasibility of implementing a BBT intervention in a military population during the high risk post-deployment window.

A sample of 74 Warriors who have deployed will be randomly placed into two groups (music with BBT and music without BBT). Each group will be exposed to their respective intervention for 30 minutes at bedtime, 3 times a week, for 4 weeks. Quantitative and qualitative measures will be collected as follows…

1. Cardiovascular reactivity, c-reactive protein, and state anxiety measures will be collected at baseline and after the 4 week intervention.
2. Morning blood pressure (BP) surge and evening BP decline measures will be collected at baseline and weeks 0, 2 and 4.
3. Input from the participants will be collected via daily logs and at the completion of the 4 week intervention.

Aim 1 - To assess the feasibility of implementing a binaural beat technology intervention in a military population during the high risk post deployment window. Feasibility will be measured by assessing:

1. retention
2. number of refusal during recruitment
3. number of drop outs
4. reason for drop outs
5. reason for staying
6. number of days the technology was used
7. selection of music
8. ease of use and comfort of equipment
9. adherence to the protocol
10. evaluation of recruitment strategies

Aim 2 - To assess the impact of binaural beat technology on anxiety and relevant CV health measures. These measures included:

1. Comparison of pre and post intervention state anxiety scores
2. Observing the trend of morning blood pressure surge over time
3. Observing the trend of evening blood pressure decline over time
4. Comparison of pre and post intervention heart rate variability measures
5. Comparison of pre and post intervention c-reactive protein measures

ELIGIBILITY:
Inclusion Criteria:

* Military personnel who

  1. Have deployed
  2. Are eligible to receive healthcare at WRNMMC or FBCH
  3. Are 18 years and older
  4. Are able to commit to a 5-week study

     Exclusion Criteria:
* Military personnel who…

  1. Are taking any medication in the anti-hypertensive category
  2. Are taking any medication in the anti-anxiety category
  3. Have been diagnosed with moderate or severe traumatic brain injury
  4. Have a history of epilepsy
  5. Are taking any medication in the anti-seizure category
  6. Have hearing deficit and/or wear a hearing aide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
C-Reactive Protein | Before the intervention and again at 5 weeks
  C-reactive protein is a biomarker of the inflammatory process.
State-Trait Anxiety (STAI) | Before the intervention and again at 5 weeks
  The STAI will be used to measure overall generalized anxiety as well as current state anxiety immediately before and after the intervention. The instrument consists of 40 4-point Likert scale statements (20 related to trait anxiety and 20 related to state anxiety). Scores range from 40 to 160 with the higher score depicting a higher level of anxiety.
Morning Blood Pressure/Evening Blood Pressure Decline | Before the intervention, at 2 weeks and again at 4 weeks
  Using an ambulatory blood pressure (BP) monitor, BP measures will be taken every 60 minutes starting from two hours before bedtime and ending two hours after rising. Morning BP surge will be assessed by comparing the trend of the number of millimeters of mercury (mm Hg) the BP increased during the first two hours after rising. Evening BP decline will be assessed by comparing the trend of the percentage that the BP declined while sleep when compared the mean awake BP.
Cardiovascular Reactivity | Before the intervention and again at 5 weeks
  Continuous heart rate measures will be taken during five states: 1) at baseline, 2) during the training for a cognitive challenge, 3) during the cognitive challenge, 4) during recovery, and 5) when verbally coached to relax. When analyzed via the computer, a high variability response will indicate a healthy autonomic system whereas a low variability response will indicate evidence of chronic stress exposure.
Post Intervention Questionnaire | At 5 weeks
  The Post Intervention Questionnaire will be used to collect qualitative data (3 questions to address efficacy and 11 questions to address feasibility). This instrument will be used in conjunction with field notes during recruitment to assess: 1) retention, 2) number of refusal during recruitment, 3) number of drop outs, 4) reason for drop out, 5) reason for staying, 6) number of day the technology was used (more or less than prescribed recommendation), 7) selection of music, 8) ease of use and comfort of equipment (e.g., sleep phone, mp3 player, etc), 9) adherence to the protocol, and 10) evaluation of recruitment strategies.

CONTACTS AND LOCATIONS:
Overall Officials: MeLisa Gantt, PhD, Principal Investigator — Gantt Clinical Research Institute LLC
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia